CLINICAL TRIAL: NCT04847453
Title: A Phase 1/1a Study of Venetoclax, MLN9708 (Ixazomib Citrate) and Dexamethasone for Relapsed/Refractory Light Chain Amyloidosis
Brief Title: Venetoclax, MLN9708 (Ixazomib Citrate) and Dexamethasone for the Treatment of Relapsed or Refractory Light Chain Amyloidosis
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2021-03038; NCI-2021-03038 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PHI-124; 10440 (Other: City of Hope Comprehensive Cancer Center LAO); 10440 (Other: CTEP); UM1CA186717 (NIH)
Record Dates: First submitted 2021-04-15; First posted 2021-04-19 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Recurrent AL Amyloidosis; Refractory AL Amyloidosis
MeSH Terms: conditions — Immunoglobulin Light-chain Amyloidosis | interventions — Specimen Handling; Biopsy; Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; ixazomib; Magnetic Resonance Spectroscopy; venetoclax; X-Rays; Phantoms, Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (venetoclax, ixazomib citrate, dexamethasone) (Experimental): Patients receive venetoclax PO QD on days 1-28, ixazomib citrate PO on days 1, 8 and 15, and dexamethasone PO on days 1, 8, 15 and 22 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients may undergo x-ray imaging and abdominal ultrasound during screening. Patients undergo ECHO during screening and bone marrow biopsy and/or aspiration as well as blood sample collection throughout the study. Patients may undergo CT scans, and/or MRI, and/or PET scans and may optionally undergo urine sample collection throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration and Biopsy; Procedure: Computed Tomography; Drug: Dexamethasone; Procedure: Echocardiography Test; Drug: Ixazomib Citrate; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Procedure: Transabdominal Ultrasound; Drug: Venetoclax; Procedure: X-Ray Imaging

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood and urine specimen collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Aspiration and Biopsy — Undergo bone marrow aspiration and biopsy
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Drug: Dexamethasone — Given PO
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycadron; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decadron DP; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasone Intensol; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Dxevo; Fluorodelta; Fortecortin; Gammacorten; Hemady; Hexadecadrol; Hexadrol; LenaDex; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; TaperDex; Visumetazone; ZoDex
Procedure: Echocardiography Test — Undergo ECHO
  Other Names: EC; Echocardiography
Drug: Ixazomib Citrate — Given PO
  Other Names: MLN 9708; MLN-9708; MLN9708; Ninlaro
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Procedure: Positron Emission Tomography — Undergo PET scan
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
Procedure: Transabdominal Ultrasound — Undergo transabdominal ultrasound
  Other Names: abdominal ultrasound; TUS
Drug: Venetoclax — Given PO
  Other Names: ABT 199; ABT-0199; ABT-199; ABT199; GDC 0199; GDC-0199; GDC0199; RG7601; Venclexta; Venclyxto
Procedure: X-Ray Imaging — Undergo x-ray
  Other Names: Conventional X-Ray; Diagnostic Radiology; Medical Imaging, X-Ray; Plain film radiographs; Radiographic Imaging; Radiographic imaging procedure (procedure); Radiography; RG; Static X-Ray; X-Ray

SUMMARY:
This phase I/Ia trial finds the best dose and side effects of venetoclax given in combination with ixazomib citrate and dexamethasone in treating patients with light chain amyloidosis that has come back (relapsed) or does not respond to treatment (refractory) and who have an abnormal genetic change [translocation t(11;14)]. Venetoclax is in a class of medications called B-cell lymphoma-2 (BCL-2) inhibitors. It may stop the growth of cancer cells by blocking Bcl-2, a protein needed for cancer cell survival. Ixazomib citrate is in a class of medications called proteasome inhibitors. It works by helping to kill cancer cells. Anti-inflammatory drugs such as dexamethasone reduce inflammation by lowering the body's immune response and are used with other drugs in the treatment of some types of cancer. Combination therapy with venetoclax, ixazomib citrate and dexamethasone may be effective in treatment of relapsed or refractory light chain amyloidosis.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the safety and tolerability of venetoclax, MLN9708 (ixazomib citrate), and dexamethasone when used in combination.

II. To determine the maximum tolerated dose (MTD) and recommended phase II dose (RP2D) of venetoclax, MLN9708 (ixazomib citrate), and dexamethasone when used in combination.

SECONDARY OBJECTIVES:

I. To observe and record anti-tumor activity. II. To obtain a preliminary estimate of the anti-light chain amyloidosis (AL) activity as assessed by incidence of complete hematologic response (CR) and overall hematologic response (partial response [PR], very good partial response [VGPR], and CR).

III. To estimate the organ-specific response rates, among patients with measurable organ disease, using standard criteria.

IV. To estimate progression free survival.

EXPLORATORY OBJECTIVES:

I. To evaluate expression of BCL-2, BCL-XL, and MCL-1 on the surface of plasma cells of patients with AL.

II. To describe the immune profile in the peripheral blood of patients with AL before and during treatment with venetoclax, MLN9708 (ixazomib citrate), and dexamethasone at multiple time points.

III. To estimate hematologic response rates using mass spectrometry to detect persistence of a monoclonal protein in the serum and urine.

IV. To characterize the genotype of the CD138+ plasma cell in patients with AL and t(11;14) and compare findings to those of patients with multiple myeloma and t(11;14) as reported in prior studies.

V. To determine presence of minimal residual disease by Next Generation Sequencing (NGS) in patients achieving a hematologic CR.

OUTLINE: This is a dose-escalation study of venetoclax and ixazomib citrate.

Patients receive venetoclax orally (PO) once daily (QD) on days 1-28, ixazomib citrate PO on days 1, 8 and 15, and dexamethasone PO on days 1, 8, 15 and 22 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients may undergo x-ray imaging and abdominal ultrasound during screening. Patients undergo echocardiography (ECHO) during screening and bone marrow biopsy and/or aspiration as well as blood sample collection throughout the study. Patients may undergo computed tomography (CT) scans, and/or magnetic resonance imaging (MRI), and/or positron emission tomography (PET) scans and may optionally undergo urine sample collection throughout the study.

After completion of study treatment, patients are followed every 1-3 months until disease progression or death.

ELIGIBILITY:
Inclusion Criteria:

* Histologically-proven systemic anti-light chain amyloidosis (AL) confirmed by positive Congo red staining with green birefringence on polarized light microscopy and evidence of a measurable clonal disease that requires active treatment. An underlying plasma cell disorder can be identified by one of the following: clonal plasma cells in the bone marrow (BM), monoclonal protein in the serum or urine, or abnormal free light chain ratio. For patients who are African-American or males >= 70 years with isolated cardiac involvement, mass spectrometry must be performed to confirm subtyping
* Presence of t(11;14) by fluorescence in situ hybridization (FISH) on bone marrow biopsy, either confirmed at screening or documented with a prior biopsy
* Patient requires therapy, as determined by the treating physician, following at least one line of treatment (No limit on the number of prior treatments)
* Age >= 18 years. Because no dosing or adverse event data are currently available on the use of venetoclax in combination with MLN9708 (ixazomib citrate) and dexamethasone in patients < 18 years of age, children are excluded from this study
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,000/mcL. Screening absolute neutrophil count (ANC) should be independent of granulocyte- and granulocyte/macrophage colony stimulating factor (G-CSF and GM-CSF) support for at least 1 week and of pegylated G-CSF for at least 2 weeks
* Platelets >= 75,000/mcL. Platelet transfusions to help patients meet eligibility criteria are not allowed within 2 weeks before study enrollment
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST)(serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT)(serum glutamate pyruvate transaminase [SGPT]) =< 3 x institutional ULN
* Creatinine Calculated clearance >= 15 mL/min using Cockcroft-Gault equation
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* AL Amyloidosis Cardiac Risk stage I, II or IIIa disease based on the 2013 European Modification of the 2004 Standard Mayo Clinic Staging in patients with advanced cardiac involvement (Dispenzieri et al., 2004; Wechalekar et al., 2013)

  * Staging system defined by: NT-proBNP cut off of < 332 pg/mL and troponin I cut-off of < 0.10 ng/mL (in the absence of troponin T, troponin I >= 0.1 ng/mL can be used) as thresholds for stages I, II and III; NT-proBNP =< 8500 pg/ml for stage IIIa
  * Stage I, both under threshold;

    * Stage I: Zero markers above threshold: NT-proBNP < 332 ng/L AND troponin T (TnT) =< 0.035 ng/mL; NT-proBNP < 332 ng/L AND TnI =< 0.1 ng/mL
  * Stage II, either troponin or NT-proBNP (but not both) over threshold;

    * Stage II: One marker above threshold: NT-proBNP >= 332 ng/L OR TnT >= 0.035 ng/mL; NT-proBNP >= 332 ng/L OR TnI >= 0.1 ng/mL
  * Stage III, both over threshold;
  * Stage IIIa, both over threshold but NT-proBNP =< 8500 pg/ml

    * Stage IIIa: Two markers above threshold: NT-proBNP >= 332 ng/L BUT =< 8,500 ng/L AND TnT >= 0.035 ng/mL; NT-proBNP >= 332 ng/L BUT =< 8,500 ng/L AND TnI >= 0.1 ng/mL
    * Stage IIIb: Two markers above threshold: NT-proBNP > 8,500 ng/L AND TnT >= 0.035 ng/mL; NT-proBNP > 8,500 ng/L AND TnI >= 0.1 ng/mL
* Life expectancy >= 3 months
* Plasma cell burden =< 60%
* Absence of bone lesions and other end organ disease consistent with multiple myeloma (patients with plasma cell burden between 10 and 60% without end organ disease can be included)
* Measurable disease of AL amyloidosis as defined by at least one of the following: 1) serum or urine monoclonal protein >= 500 mg/dL by protein electrophoresis, or 2) serum free light chain >= 20 mg/L with an abnormal kappa:lambda ratio or the difference between involved and uninvolved free light chains (dFLC) >= 20 mg/L
* It is not known what effects MLN9708 (ixazomib citrate), venetoclax, and dexamethasone have on human pregnancy or development of the embryo or fetus. Therefore, female patients participating in this study should avoid becoming pregnant, and male patients should avoid impregnating a female partner. Nonsterilized female patients of reproductive age group and male patients should use effective methods of contraception through defined periods during and after study treatment as specified below.

  * Female patients must meet 1 of the following:

    * Postmenopausal for at least 1 year before the screening visit, or
    * Surgically sterile, or
    * If they are of childbearing potential, agree to practice 2 effective methods of contraception from the time of signing of the informed consent form through 90 days after the last dose of study drug, or
    * Agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [e.g., calendar, ovulation, symptothermal, postovulation methods] and withdrawal are not acceptable methods of contraception)
  * Male patients, even if surgically sterilized (i.e., status postvasectomy) must agree to 1 of the following:

    * Practice effective barrier contraception during the entire study treatment period and through 90 days after the last dose of study drug, or
    * Agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [e.g., calendar, ovulation, symptothermal, postovulation methods for the female partner] and withdrawal are not acceptable methods of contraception)
* Left ventricular ejection fraction >= 35% by echocardiogram.
* Ability to understand and the willingness to sign a written informed consent document. Participants with impaired decision-making capacity (IDMC) who have a legally-authorized representative (LAR) and/or family member available will also be eligible

Exclusion Criteria:

* Patients who have had major surgery or radiotherapy within 14 days prior to entering the study. If the involved radiotherapy field is small, 7 days will be considered a sufficient interval between treatment and administration of the MLN9708 (ixazomib citrate)
* Patients who have had anti-plasma cell therapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study
* Patients who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > grade 1) with the exception of alopecia
* Patients who are receiving any other investigational agents, within 30 days of the start of this trial and throughout the duration of this trial
* Patients with central nervous system involvement
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to venetoclax, MLN9708 (ixazomib citrate) (including boron or boron-containing products) or dexamethasone
* Strong or moderate CYP3A inhibitors (e.g., erythromycin, ciprofloxacin, diltiazem, fluconazole, verapamil), or strong CYP3A inducers (e.g., carbamazepine, phenytoin, rifampin, St. John's wort), or moderate CYP3A inducers (e.g., bosentan, efavirenz, etravirine) should be avoided
* Venetoclax should be administered using caution with substrates or inhibitors of P-glycoprotein (P-gp)
* Patients with uncontrolled intercurrent illness including, but not limited to: ongoing or active serious or systemic infection (within 14 days prior to study enrollment), active hepatitis B or C virus infection, hypertension, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or myocardial infarction (within the past 6 months)
* Patients with psychiatric illness/social situations that would limit compliance with study requirements
* Female patients who are lactating or have a positive serum pregnancy test during the screening period are excluded from this study because MLN9708 (ixazomib citrate) is a proteasome inhibitor with the potential for embryo-lethal effects, and an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with MLN9708 (ixazomib citrate). Patients must stop breastfeeding while on MLN9708 (ixazomib citrate) and until 90 days have passed since their last dose. These potential risks may also apply to other agents used in this study
* Known gastrointestinal disease or gastrointestinal procedure that could interfere with the oral absorption or tolerance of MLN9708 (ixazomib citrate), including difficulty swallowing
* Peripheral neuropathy that is >= grade 3, or grade 2 with pain on clinical examination during the screening period
* Patients that have previously been treated with MLN9708 (ixazomib citrate). Patients who have received prior treatment with venetoclax
* Patients without measurable disease by serum free light chain, serum m-spike or urine monoclonal protein
* Patients with New York Heart Association classification III/IV. Patients with advanced cardiac amyloidosis, Mayo stage IIIB based on European Modification of the 2004 Standard Mayo Clinic Staging in patients with advanced cardiac involvement with NT-Pro BNP > 8500 pg/mL (Wechalekar et al., 2013)
* Patients with grade 3 or worse diarrhea

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-08-03 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 30 days
  Toxicity will be evaluated according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0.
Maximum tolerated dose | Up to the end of cycle 1
  Defined as the dose for which the isotonic estimate of the toxicity rate is closest to the target toxicity rate.
Recommended phase 2 dose (RP2D) | Up to the end of cycle 1
  Will be based on the assessment of toxicities during cycle 1 that meet criteria for dose-limiting toxicities (DLT).

SECONDARY OUTCOMES:
Overall response rate (complete hematologic response) | After cycles 3, 6, 9, and 12, and every 6 months thereafter up to 2.5 years
  Will be estimated based on the patients enrolled in the dose-escalation as well as the dose-expansion stage, using Clopper-Pearson confidence interval. Hematologic complete response rate will be evaluated according to the consensus guidelines in treatment response.

OTHER OUTCOMES:
Expression of BCL-2, BCL-XL, BAX, BAK, BIM, NOXA, and MCL-1 | Baseline
  Will be assessed by immunohistochemistry.
Immune profile in the peripheral blood | Before and during treatment
  Will be determined by mass cytometry.
Hematologic response rates | Up to 2.5 years
  Estimated using mass spectrometry to detect persistence of a monoclonal protein in the serum and urine.
Characterization of CD138+ plasma cell with t(11;14) | Up to 2.5 years
Presence of minimal residual disease | Up to 2.5 years
  Will be determined by Next Generation Sequencing in patients achieving a hematologic complete response.

CONTACTS AND LOCATIONS:
Overall Officials: Michael A Rosenzweig, Principal Investigator — City of Hope Comprehensive Cancer Center LAO
Locations (16):
- United States (16):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - University of Texas at Austin, Austin, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm

REFERENCES:
- [Derived] Locke M, Nieto M. AL Amyloidosis: Current Treatment and Outcomes. Adv Hematol. 2025 Mar 3;2025:7280805. doi: 10.1155/ah/7280805. eCollection 2025. PMID 40226119